CLINICAL TRIAL: NCT07377578
Title: A Randomized, Open-label, Multicenter, Phase III Clinical Study Comparing Rocbrutinib Monotherapy Versus Investigator's Choice of BTK Inhibitors in Patients With Relapsed or Refractory Mantle Cell Lymphoma (MCL) (PRIME Study)
Brief Title: A Study of Rocbrutinib Versus Investigator's Choice of BTK Inhibitors in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP-168-CN302
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; BTK inhibitor; Rocbrutinib
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; acalabrutinib; zanubrutinib; orelabrutinib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Rocbrutinib) (Experimental)
  Interventions: Drug: Rocbrutinib
- Arm B (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib) (Active Comparator)
  Interventions: Drug: Ibrutinib; Drug: Acalabrutinib; Drug: Zanubrutinib; Drug: Orelabrutinib

INTERVENTIONS:
Drug: Rocbrutinib — Rocbrutinib at 150 mg once daily orally until disease progression or unacceptable toxicity
  Arms: Arm A (Rocbrutinib)
Drug: Ibrutinib — Ibrutinib, 560 mg once daily orally and continuously
  Arms: Arm B (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib)
Drug: Acalabrutinib — Acalabrutinib, 100 mg twice daily orally and continuously
  Arms: Arm B (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib)
Drug: Zanubrutinib — Zanubrutinib, 160 mg twice daily orally and continuously
  Arms: Arm B (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib)
Drug: Orelabrutinib — Orelabrutinib, 150 mg once daily orally and continuously
  Arms: Arm B (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib)

SUMMARY:
Mantle cell lymphoma (MCL) is an aggressive yet often indolent type of B-cell non-Hodgkin lymphoma (NHL). Rocbrutinib (LP-168) is a novel, highly selective, fourth-generation Bruton's tyrosine kinase (BTK) inhibitor that exhibits both covalent (irreversible) and non-covalent (reversible) binding. This unique dual mechanism of action has shown promising efficacy and a favorable safety profile across various B-cell NHL subtypes in prior Phase 1 and 2 studies. This is a Phase 3, randomized, open-label study comparing Rocbrutinib versus investigator's choice of BTK inhibitor (ibrutinib, acalabrutinib, zanubrutinib, or orelabrutinib) in patients with MCL who have received at least one prior line of therapy and are naïve to BTK inhibitor treatment (except for intolerance).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MCL, who have received at least one prior systemic regimen(s), and have experienced disease progression on the most recent line of therapy.
* Have at least one measurable lesion according to the Lugano Response Criteria 2014.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2.
* Life expectancy ≥ 12 weeks.
* Adequate coagulation function, liver and kidney function, bone marrow hematopoietic function, etc.
* Toxicities or complications from prior anti-tumor therapy have recovered to Grade ≤1 according to NCI CTCAE v5.0.
* All male subjects and female subjects of childbearing potential must strictly use medically approved contraception throughout the entire study period. All male subjects must also avoid sperm donation during the above period. For women of childbearing potential, the result of serum pregnancy test must be obtained. Women must be non-lactating.
* Subject voluntarily enrolls and signs the informed consent form, and agrees to comply with the study treatment plan and visit schedule.

Exclusion Criteria:

* Hypersensitivity to Rocbrutinib or any study drug in the control group.
* Prior treatment with any BTK-targeted therapy (except for intolerance).
* Central nervous system (CNS) involvement by lymphoma.
* History of other malignancy (except MCL) within the past 2 years, excluding radically cured skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ, localized squamous cell carcinoma, etc.
* History of major cardiovascular events within 6 months prior to randomization.
* Presence of any severe and/or uncontrolled systemic disease that, in the investigator's judgment, or have poor cardiac function.
* Uncontrolled active bacterial, fungal, or viral systemic infection, or active tuberculosis infection.
* Any medical condition that could interfere with the absorption, distribution, metabolism, or excretion (ADME) of the investigational drug or the evaluation of study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2031-05-30 (Estimated); Study Completion 2033-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by IRC | approximately 30 months

SECONDARY OUTCOMES:
PFS assessed by INV | approximately 30 months
Overall Response Rate (ORR) assessed by IRC and INV, respectively | Up to approximately 24 months
Duration of Response (DOR) assessed by IRC and INV, respectively | approximately 30 months
Overall Survival | approximately 40 months
Number of participants with treatment-emergent adverse event as assessed by CTCAE v5.0 | Up to approximately 40 months
Number of participants with treatment-related adverse event as assessed by CTCAE v5.0 | Up to approximately 40 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: No